CLINICAL TRIAL: NCT06783660
Title: A Multicenter, Open-label, Randomized, Independent Evaluation, Confirmatory Clinical Trial to Evaluate the Safety and Efficacy of the Periodontal Tissue Inducing Photoresponsive PeptiCol EZgraft in the Extraction Socket Preservation Process After Tooth Extraction.
Brief Title: PeptiCol EZgraft in the Extraction Socket Preservation Process After Tooth Extraction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NIBEC Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIB-IND-(PTC)CTP; RS-2020-KD000091 (Other Grant/Funding Number: The Korea Medical Device Development Fund)
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-01

CONDITIONS: Alveolar Ridge Augmentation
Keywords: socket preservation; collagen sponge; collagen gel; Peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peptide-loaded collagen sponge and collagen gel complex (Experimental): A piece of peptide-loaded collagen sponge (Regenomer®) was placed in an extraction socket after tooth extraction and cover wound with collagen gel.
  Interventions: Device: Peptide-loaded collagen sponge and collagen gel complex
- Collagen sponge (Active Comparator): A piece of collagen sponge（Regenomer®）was placed in an extraction socket after tooth extraction.
  Interventions: Device: Collagen sponge

INTERVENTIONS:
Device: Peptide-loaded collagen sponge and collagen gel complex — A piece of peptide-loaded collagen sponge (Regenomer®) and collagen gel complex
  Arms: Peptide-loaded collagen sponge and collagen gel complex
Device: Collagen sponge — Type 1 Collagen sponge (Regenomer)
  Arms: Collagen sponge

SUMMARY:
This clinical trial aims to compare the efficacy and safety of applying "PeptiCol EZgraft" in extraction socket preservation procedures against "Regenomer," in terms of reducing the amount of alveolar bone change during the healing process following tooth extraction.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to compare the efficacy and safety of using "PeptiCol EZgraft" in extraction socket preservation procedures against "Regenomer," specifically to evaluate whether PeptiCol EZgraft is more effective in reducing alveolar bone changes compared to Regenomer. The trial aims to assess both the effectiveness and safety of PeptiCol EZgraft in minimizing alveolar bone resorption during the healing process following tooth extraction.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 to 75 years.
2. Systemically healthy or with mild systemic disease, classified as ASA I or II.
3. Planning to place implants in the maxilla or mandible after extraction, or having such plans for the future. If there are multiple extraction sockets, only one socket will be included in the trial, and other areas will follow spontaneous healing or treatment plans.
4. The extraction socket area must have more than 50% of the alveolar bone wall remaining.
5. Willing to maintain good oral hygiene during the clinical trial.
6. Voluntarily decided to participate in the trial and signed the informed consent form.
7. Willing to participate for the entire duration of the clinical trial and comply with trial procedures.

Exclusion Criteria:

1. Extensive alveolar bone absorption observed in the extraction socket area.
2. Severe periodontal disease or acute periodontal abscess.
3. Poor oral hygiene.
4. History of bone grafts or implants in the area of the medical device application.
5. Mucosal diseases due to autoimmune disorders.
6. History of hypersensitivity to collagen preparations.
7. Smoking more than 10 cigarettes per day.
8. Alcohol or drug addiction.

   *The alcohol addiction screening will be conducted using AUDIT-K.
9. Use of drugs affecting bone formation within 2 weeks prior to screening (e.g., steroids, bisphosphonates).
10. Use of oral or injectable rheumatic medications, including immunosuppressants, within 2 weeks prior to screening.
11. History of or current use of oral or injectable bisphosphonates for osteoporosis for more than 12 weeks.
12. Uncontrolled bleeding disorders or use of medications affecting blood coagulation.
13. Uncontrolled diabetes or hypertension.
14. Clinically significant cardiovascular, gastrointestinal, respiratory, endocrine, or central nervous system diseases observed at screening.
15. Immune disorders including acquired immunodeficiency syndrome.
16. Pregnant or breastfeeding women
17. During the clinical trial period, female and male participants who are of childbearing potential must agree to use appropriate contraception from the date of signing the informed consent form until the end of the clinical trial (16 weeks post-procedure). If a female participant becomes pregnant during the trial period, her participation will be discontinued.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Measure the change in alveolar bone width at the 25% point of the extraction socket on CBCT images at 4 months compared to baseline | at 4 months compared to baseline
  To apply reproducible endpoints, a reference stent, was placed in the oral cavity before the procedure and CBCT images were taken at baseline and 4 months after the test/control device was placed to assess the change in alveolar bone width at the upper 25% of the alveolar bone between the test and control groups.
Evaluation of safety measures via occurrence of (S)AE ((serious) adverse events), DD (device deficiency) and medical device related events | 4 months, evaluation at each visit
  * List all anticipated side effects and adverse events with detailed descriptions.
    * Record the frequency of adverse events related and unrelated to the clinical trial device.
      * List all adverse events with detailed descriptions and record the frequency of events related and unrelated to the clinical trial device.
        * Compare the number of adverse events related to the clinical trial device across treatment groups.
          * Compare the number of adverse events related to the clinical trial medical device by each treatment group.

SECONDARY OUTCOMES:
Participant satisfaction evaluation | at 4 months compared to baseline
  Participant evaluations such as satisfaction with the procedure and pain assessment were collected after the procedure. A survey was conducted using a 5-point scale from "very dissatisfied to very satisfied"
Assessment of alveolar bone healing | at 4 months compared to baseline
  The goal is to measure the variables to observe the healing of alveolar bone based on CBCT at 4 months from baseline.
  1. Change in bone width Bone width at 50 and 75% of the alveolar bone apex at baseline and at 4 months with the investigational/control device was measured using CBCT scans taken with the reference stent in the oral cavity.
  2. Change in bone height D2 measured from line C as described by Fiorellini et al. at baseline to line C at 4 months after application of the test/control device, using CBCT images taken with the reference stent in the oral cavity.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Dental Hospital, Korea, Seoul, South Korea